CLINICAL TRIAL: NCT05994469
Title: Prevention of Groin Injuries in Rink Hockey: A One Season Natural Experiment
Brief Title: Prevention of Groin Injuries in Rink Hockey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Principal Investigator, University of Oviedo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UO2023/1
Record Dates: First submitted 2023-08-05; First posted 2023-08-16 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Groin Injury; Groin Strain; Adductor Strain
Keywords: rink hockey; groin pain; injury prevention

STUDY DESIGN:
Intervention Model Description: Natural experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copenhagen Adduction Exercise Group (Experimental): there is no control group, all teams can implement the intervention protocol that better fits their normal schedule, the intervention can consist of 1 or 2 Copenhagen Adduction Exercise sessions per week
  Interventions: Behavioral: Copenhagen Adduction Exercise

INTERVENTIONS:
Behavioral: Copenhagen Adduction Exercise — The CAE is performed by side-lying on the floor with the dominant lower limb supported in the air by a teammate, the hip is adducted until the body forms a straight line from the ankles to the shoulders (concentric phase), then the player is instructed to lower the body slowly (eccentric phase) until reaching the floor to start the next repetition.

SUMMARY:
Rink hockey teams from senior category (adults) will be recruited to implement a groin injury prevention program consisting on the Copenhagen Adduction Exercise (CAE) throughout the regular season, 0 times, once or twice per week (september 2023-march 2024)

Weekly team exposure to training sessions and games will be collected as well as cases of groin problems in the entire population

When the season ends, the number of groin problems will be compared between teams that used the prevention program once a week against twice a week or no sessions a week.

DETAILED DESCRIPTION:
Rink hockey teams will be offered a prevention program consisting on the CAE to be performed during the season.

Teams will decide to implement the protocol once, twice or 0 times per week, depending on their schedule. No formal control group will be set, comparison of injuries will be performed between teams that used +80% of the total possible sessions and -80% (28 weeks equals a potential 42 CAE sessions throughout the season).

On a weekly basis, coaches will be contacted to report number of training sessions, games, and training sessions where they implemented CAE.

Bi-weekly, players will report any episode of groin problems (both leading to time-loss and those only affecting performance while not limiting participation).

ELIGIBILITY:
Inclusion Criteria:

* #1 Be part of a rink hockey team competing in senior league (either local (third division/lower) or national (first and second division))

  * 2 Accept participating in the study (signing the informed consent)

Exclusion Criteria:

* #1 not playing rink hockey in the previous season

  * 2 serious illness, injury or surgery in the previous 6 months that prevented rink hockey participation

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Bi-Weekly prevalence of groin problems | Every 14 days throughout the entire study (which lasts 7 months)
  number of groin pain complaints in a 14-day frame, groin pain is described as pain in the groin region which emerges from performing exercise and may be indicative of an injury to the adductor muscles, abdominals, hip flexors, or pubic joint

SECONDARY OUTCOMES:
Adherence to the intervention | Every 7 days throughout the entire study (which lasts 7 months)
  Since the intervention is implemented on a weekly basis, the number of sessions performed by the participating teams will be collected to calculate the total compliance with the intervention. From a total of 56 possible sessions a team may complete 47 which equals 83% compliance
hockey exposure | Every 7 days throughout the entire study (which lasts 7 months)
  number of training sessions and games per week this metric is collected to calculate exposure hours, so that groin problems can be compared as nº of injuries / 1000 hours of exposure, as the International Olympic Committee recommends

CONTACTS AND LOCATIONS:
Locations (1):
- Hugo Olmedillas, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Previous research similar to this project — https://pubmed.ncbi.nlm.nih.gov/29891614/
- See also: Previous research similar to this project — https://doi.org/10.1007/s00167-021-06644-2